CLINICAL TRIAL: NCT05421013
Title: An Open Label, Dose Escalation Study to Evaluate the Safety and Efficacy of Intralesional Injection of STP705 in Adult Subjects With Facial Cutaneous Squamous Cell Carcinoma in Situ (isSCC)
Brief Title: Study to Evaluate Safety, Efficacy of Intralesional Injection of STP705 in Adults With Facial isSCC
Acronym: isSCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-705-011
Record Dates: First submitted 2022-06-12; First posted 2022-06-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Facial isSCC
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: 3 cohorts. In the absence of DLT, subsequent cohorts will receive increasing dose of STP705
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- STP705 30ug (Experimental): STP705 will be administered once weekly for 6 weeks
  Interventions: Drug: STP705
- STP705 60ug (Experimental): STP705 will be administered once weekly for 6 weeks
  Interventions: Drug: STP705
- STP705 90ug (Experimental): STP705 will be administered once weekly for 6 weeks
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — STP705 targets TGFB-1 and COX-2 mRNA respectively.
  Other Names: STP705 Powder for Injection

SUMMARY:
Open label, dose escalation to evaluate safety.

DETAILED DESCRIPTION:
Evaluate safety, tolerability, and efficacy of various doses of STP705 administered as intralesional injection in subjects with facial isSCC.

There will be 3 cohorts of 10 subjects each. Enrolled subjects will receive STP705 once weekly for 6 weeks. The lesion will be excised 60 days after.

ELIGIBILITY:
INCLUSION CRITERIA

Inclusion Criteria: Subjects are required to meet all of the following criteria for enrollment into the study:

1. Male or female adult ≥ 18 years of age.
2. Primary, histologically confirmed facial isSCC lesion suitable for excision with a minimum diameter of 0.5 cm and with a maximum diameter of 2.0 cm.
3. Histological diagnosis of a qualified isSCC skin lesion (evidenced by a confirmatory histopathology report) made no more than 6 months prior to the screening visit.
4. No other dermatological disease in the isSCC target lesion or surrounding area, which in the opinion of the investigator, could interfere with the study.
5. Willing to refrain from using non-approved lotions or creams on the target lesion and surrounding area during the treatment period (sunscreen and moisturizers allowed).
6. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study.
7. Laboratory values for the tests (listed in the Study Schedule) within the reference ranges as defined by the local laboratory, or "out of range" test results that are clinically acceptable to the investigator.
8. Ability to follow study instructions and likely to complete all study requirements.
9. Written informed consent obtained, including consent for tissue to be examined and stored by the Central Histology Lab.
10. Written consent to allow photographs of the target isSCC lesion to be used as part of the study data and documentation.
11. For female subjects of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral / implantable / injectable / transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy at least 6 months prior to screening).

EXCLUSION CRITERIA

1. Pregnant, lactating, or planning to become pregnant.
2. Presence of known or suspected systemic cancer.
3. Confirmatory histological report of the qualified isSCC lesion reveals evidence of severe squamous metaplasia, infiltrative, desmoplastic or micronodular growth patterns in the opinion of the investigator.
4. History of recurrence of the target isSCC lesion.
5. Concurrent disease or treatment that suppresses the immune system.
6. Subjects with baseline QT corrected interval QTc > 480 msec using Fridericia's formula.
7. Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk.
8. Known sensitivity to any of the ingredients in the study medication including an allergy to trehalose.
9. Use of a tanning bed or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the study.
10. Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit.
11. Use of systemic retinoids within the 6 months prior to the screening period.
12. Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period.
13. Use of topical immunomodulators within 2 cm of the target isSCC lesion within the 4 weeks prior to the screening period.
14. Treatment with the following topical agents within 2 cm of the target isSCC lesion within the 4 weeks prior to the screening visit: aminolevulinic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, ingenol mebutate, tirbanibulin, or imiquimod.
15. Treatment with liquid nitrogen, surgical excision, or curettage within 2 cm of the target isSCC lesion during the 4 weeks prior to the screening visit.
16. Evidence of current chronic alcohol or drug abuse that, in the opinion of the investigator, would impair the subject's ability to comply with study schedule.
17. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit.
18. In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with histological clerance of treated isSCC lesion at the end of treatment | 21 weeks
  Histological clearance will be defined as the absence of detectable evidence of isSCC tumor cell nests determined by pathology review

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 21 weeks
  The following Treatment Emergent AEs (TEAEs): System organ Class and preferred term will be coded using Medical Dictionary for Regulatory Activities (MedDRA):
  Overall: (regardless of severity or relationship to treatment) Intensity: (mild, moderate, severe, life threatening) Causality: (definitely, probably, possible, likely, unrelated) Impact on study treatment (dose increased, dose not changed, dose rate reduced, dose reduced, drug interrupted, drug withdrawn, not applicable, unknown)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States